CLINICAL TRIAL: NCT05671601
Title: Application of Deep Learning Automation Based on Time-lapse Imaging to Jointly Assess Embryo Development to Improve Pregnancy Outcome of Single Blastocyst Transfer
Brief Title: Application of Deep Learning to Jointly Assess Embryo Development to Improve Pregnancy Outcome of Embryo Transfer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: wangshanshan820
Record Dates: First submitted 2022-12-05; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-11

CONDITIONS: Reproductive Medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- TLI+AI Assessment Group
  Interventions: Diagnostic Test: Automatic picture recognition
- Morphological Assessment Group
  Interventions: Diagnostic Test: Manual Assessment Group

INTERVENTIONS:
Diagnostic Test: Automatic picture recognition — A machine that processes photographs automatically taken
  Groups: TLI+AI Assessment Group
Diagnostic Test: Manual Assessment Group — Manual recognition of pictures
  Groups: Morphological Assessment Group

SUMMARY:
Aim of this research is to apply the deep learning automation based on Time-lapse imaging to jointly assess embryo development，so that it can ensure the consistency of embryo evaluation and improve the accuracy of evaluation.

DETAILED DESCRIPTION:
This study is an observational prospective study after a retrospective analysis. It is a single-center study without randomization or blindness. In the early stage, 1000 patients are collected from three periods of embryo culture through Time-lapse to establish an automated joint evaluation system for the whole process of embryo development. At the later stage, the patients are divided into two groups: Time-Lapse imaging (TLI) +Artificial Intelligence(AI) assessment group and morphological assessment group. 100 patients with Day 5 single blastocyst transplantation are carried out to follow up the pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age < 40 years old; (2) Routine IVF cycles; (3) Period number ≤ 2; (4) The number of ova collected is 5-15; (5) BMI: 18-25 kg/m 2, follicle stimulating hormone(FSH) ≤ 12 IU/L on the third day; (6) Patients with more than 3 high-quality embryos on Day3 and performed single blastocyst transplantation on day 5. (7) Patient without endometrial factors.

Exclusion Criteria:

* (1) Preimplantation Genetic Testing(PGT) is needed due to male infertility, ovulation cycle and chromosome abnormalities; (2) there are systemic diseases of clinical significance; (3) Pictures of blastocysts are not formed or available; (4) Incomplete or unclear image collection in prokaryotic, mitotic and blastocyst phases affected AI evaluation.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients are under 40 years old and need artificial intervention to have children
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
implantation rate | 2022-2023
  the probability of successful implantation of the embryo into the uterus

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05671601/Prot_000.pdf
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05671601/ICF_001.pdf